CLINICAL TRIAL: NCT00004310
Title: Phase II Randomized Study of Intravenous Versus Oral Clomipramine in Patients With Obsessive Compulsive Disorder
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Stanford University (Other)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11812; SUMC-36784
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: anxiety disorder; disease-related problem/condition; neurologic and psychiatric disorders; obsessive compulsive disorder; oncologic disorders; rare disease
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Clomipramine

INTERVENTIONS:
Drug: Clomipramine

SUMMARY:
OBJECTIVES:

I. Evaluate the efficacy of intravenous versus oral pulse loading of clomipramine (CMI) followed by a 12-week course of maintenance therapy in patients with obsessive compulsive disorder.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, multicenter study. Patients are stratified by participating institution. Patients are randomized into one of two treatment arms.

Arm I: Patients receive a pulse loading dose of clomipramine (CMI) IV and an oral placebo on days 1 and 2.

Arm II: Patients receive an oral pulse loading dose of CMI and an IV placebo on days 1 and 2.

Patients receive maintenance therapy with daily oral CMI for 12 weeks beginning 4 days after pulse loading.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Primary diagnosis of obsessive compulsive disorder (OCD) for at least 1 year Meets Diagnostic and Statistical Manual (DSM-IV) criteria by structured clinical interview Yale-Brown Obsessive-Compulsive Scale (YBOCS) score at least 20 At least 12 if only obsessions or compulsions present Secondary diagnosis of major depression eligible if: Meets DSM-IV criteria Onset occurs after OCD OCD is primary diagnosis and dominates clinical picture Excluded diagnoses: Organic mental disorder Principal psychiatric disorder other than OCD Bipolar disorder Schizophrenia Post-traumatic stress disorder Tics or Tourette's syndrome Body dysmorphic disorder Delusional disorder Borderline or schizotypal personality disorder Anorexia nervosa Bulimia nervosa Panic disorder Panic attacks Must have failed at least 2 prior regimens of serotonin re-uptake inhibitor therapy --Prior/Concurrent Therapy-- Endocrine therapy: Concurrent thyroid medication allowed if stable at least 3 months At least 2 weeks since prior systemic corticosteroids Surgery: No prior psychosurgery or other neurosurgery Other: At least 3 months since prior electroconvulsive or insulin shock therapy At least 6 weeks since prior fluoxetine At least 30 days since prior investigational drugs At least 2 weeks since any of the following: Neuroleptics (6 weeks since depot neuroleptics) Nondepot antipsychotics Anxiolytics Stimulants Barbiturates Antidepressants (4 weeks since monoamine oxidase inhibitors) At least 2 weeks since prior anticonvulsants No concurrent antipsychotics No concurrent antihypertensives, e.g., guanethidine or clonidine No concurrent behavior therapy --Patient Characteristics-- Hematopoietic: No anemia No drug-induced leukopenia No bleeding disorder No other blood dyscrasia or bone marrow depression Hepatic: Liver function tests no greater than twice normal No hepatic abnormality Renal: No renal abnormality, e.g., urinary retention Cardiovascular: No cardiac abnormality, e.g.: Congestive heart failure Myocardial infarction Cardiac conduction disturbance other than first-degree heart block Electrocardiogram with significant abnormality No hypertension Pulmonary: No pulmonary abnormality Other: No hypersensitivity to or prior severe adverse experience with clomipramine No medical contraindication to serotonin re-uptake inhibitors or tricyclic antidepressants No history of seizures and not at risk of seizures, i.e.: No family history of epilepsy No birth trauma No significant head trauma No meningitis or encephalitis No subarachnoid hemorrhage No episodes of unconsciousness, including syncope No prostatic hypertrophy No narrow-angle glaucoma, i.e., intraocular pressure greater than 22 mm Hg No uncontrolled hyperthyroidism No other clinically significant abnormality, e.g.: Neurologic Metabolic Gastrointestinal Autoimmune No substantial risk of suicide At least 6 months since drug or alcohol abuse or dependence No illiteracy No Intelligence Quotient below 80 No plan for blood donation during study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76
Dates: Start 1999-10

CONTACTS AND LOCATIONS:
Overall Officials: Lorrin Koran, Study Chair — Stanford University
Locations (2):
- United States (2):
  - Stanford University Medical Center, Stanford, California
  - University of Cincinnati Medical Center, Cincinnati, Ohio

REFERENCES:
- [Background] Koran LM, Sallee FR, Pallanti S. Rapid benefit of intravenous pulse loading of clomipramine in obsessive-compulsive disorder. Am J Psychiatry. 1997 Mar;154(3):396-401. doi: 10.1176/ajp.154.3.396. PMID 9054789